CLINICAL TRIAL: NCT01335594
Title: Clinical, Endoscopical and Manometric Evaluation of Swallowing in Obstructive Sleep Apnea Syndrome
Brief Title: Evaluation of Swallowing in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luciana Almeida Moreira da Paz Oliveira (Other)
Responsible Party: Sponsor-Investigator, Luciana Almeida Moreira da Paz Oliveira, physician, Hospital do Servidor Publico Estadual
Organization: Hospital do Servidor Publico Estadual (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SAOS2011
Record Dates: First submitted 2011-04-11; First posted 2011-04-14 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep apnea, obstructive; Deglutition Disorders; Manometry; Endoscopy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: clinical, endoscopical and manometric evaluation — clinical evaluation: questionnaire endoscopical analysis manometry

SUMMARY:
The purpose of this study is to test the hypothesis that obstructive sleep apnea syndrome is associated with deviant pharyngeal swallowing function, using clinical, endoscopical and manometric evaluation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of obstructive sleep apnea syndrome

Exclusion Criteria:

* other causes of dysphagia
* pharyngeal surgery
* prior treatment for obstructive sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of swallowing in obstructive sleep apnea | within the first 3 months after diagnostic

SECONDARY OUTCOMES:
Manometric evaluation of swallowing in obstructive sleep apnea | within the first 3 months after diagnostic
Endoscopic evaluation of swallowing in obstructive sleep apnea | within the first 3 months after diagnostic

CONTACTS AND LOCATIONS:
Overall Officials: Luciana A M da Paz Oliveira, Principal Investigator — Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo
Locations (1):
- Instituto de Assistência Médica ao Servidor Público Estadual, São Paulo, São Paulo, Brazil